CLINICAL TRIAL: NCT05950945
Title: A Phase 3b, Multicenter, Global, Interventional, Open-label Study of Trastuzumab Deruxtecan (T-DXd), an Anti-HER2-Antibody Drug Conjugate (ADC), in Subjects Who Have Unresectable and/or Metastatic HER2-low or HER2 Immunohistochemistry (IHC) 0 Breast Cancer (DESTINY-Breast15)
Brief Title: Trastuzumab Deruxtecan (T-DXd) in Patients Who Have Hormone Receptor-negative and Hormone Receptor-positive HER2-low or HER2 IHC 0 Metastatic Breast Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DS8201-0001-CIS-MA; 2023-505616-38-00 (Other: EU CT)
Record Dates: First submitted 2023-05-22; First posted 2023-07-18 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Breast Cancer
Keywords: Trastuzumab Derextecan; Enhertu®; DS8201-a; Breast Cancer; Anti-HER2-Antibody Drug Conjugate
MeSH Terms: conditions — Breast Neoplasms | interventions — trastuzumab deruxtecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1: HR-negative, HER2-low (Experimental): Participants with HR-negative HER2-low unresectable and/or metastatic breast cancer who have received at least one and at most two prior lines of therapy in the metastatic setting will receive T-DXd.
  Interventions: Drug: Trastuzumab Deruxtecan
- Cohort 2: HR-negative, HER2 IHC 0 (Experimental): Participants with HR-negative HER2 IHC 0 unresectable and/or metastatic breast cancer who have received at least one and at most two prior lines of therapy in the metastatic setting will receive T-DXd.
  Interventions: Drug: Trastuzumab Deruxtecan
- Cohort 3: HR-positive, HER2-low (Experimental): Participants with HR-positive HER2-low unresectable and/or metastatic breast cancer who have received at least one and at most two prior lines of therapy in the metastatic setting will receive T-DXd.
  Participants must also have recurrent disease <2 years from the initiation of adjuvant ET or have disease progression on CDK4/6 inhibitor-based regimen within 12 months of completion of adjuvant therapy with a CDK4/6 inhibitor or have disease progression within the first 12 months of CDK4/6 in the first line metastatic setting.
  Interventions: Drug: Trastuzumab Deruxtecan
- Cohort 4: HR-positive, HER2 IHC 0 (Experimental): Participants with HR-positive HER2 IHC 0 unresectable and/or metastatic breast cancer who have received at least one and at most two prior lines of therapy in the metastatic setting will receive T-DXd.
  Interventions: Drug: Trastuzumab Deruxtecan

INTERVENTIONS:
Drug: Trastuzumab Deruxtecan — Intravenous administration, 5.4 mg/kg on Day 1 of each 21-day cycle until radiographic disease progression as assessed by the investigator, unacceptable toxicity, other discontinuation criteria are met, or 2 years after first dose of study drug
  Other Names: T-DXd; DS-8201a (trastuzumab derextecan); Enhertu®

SUMMARY:
This study will evaluate the safety and efficacy of trastuzumab deruxtecan (T-DXd) in participants with human epidermal growth factor receptor 2 (HER2)-low or HER2 immunohistochemistry (IHC) 0 (who are both hormone receptor [HR]-negative and HR-positive) unresectable and/or metastatic breast cancer.

DETAILED DESCRIPTION:
The primary endpoint of interest in this study is time to next treatment (TTNT), a measure that will determine how long T-DXd allows patients to derive clinical benefit from the study drug.

ELIGIBILITY:
Inclusion Criteria:

* Sign and date the main informed consent form
* Must agree to provide a newly obtained or archival baseline biopsy from primary and/or metastatic lesion.
* Pathologically documented Breast Cancer (BC) tumor

  * Is unresectable and/or metastatic.
  * Is hormone receptor-negative or hormone receptor-positive.

    * Must include percentage of positively stained cells to characterize if hormone receptor-positive or -negative.
  * Has confirmed HER2 IHC 1+ or IHC 2+/ISH- (HER2-low) status or HER2 IHC 0 status as determined according to ASCO CAP 2018 guidelines1 based on sample collected during Tissue Screening as described above.
  * Was never previously HER2-positive (IHC 3+ or IHC 2+/ISH+) on prior pathology testing (per ASCO CAP guidelines).
  * Was never previously treated with anti-HER2 therapy in the metastatic setting.
* Has had at least one and up to two prior lines of therapy in the metastatic setting.

  * In participants with hormone receptor-positive HER2-low metastatic BC (Cohort 3):

    * Has recurrent disease <2 years from the initiation of adjuvant ET OR
    * Has disease progression on CDK4/6 inhibitor-based regimen within 12 months of completion of adjuvant therapy with a CDK4/6 inhibitor OR
    * Has disease progression within the first 12 months of CDK4/6 in the first line metastatic setting
* Presence of at least one measurable lesion based on computed tomography or magnetic resonance imaging.
* Participants with brain metastases are allowed in the study. The brain lesion(s) should be small (<2 cm), untreated, asymptomatic, not requiring urgent medical intervention, and are asymptomatic and clinically stable.
* Has an Eastern Cooperative Oncology Group performance status of 0 or 1.
* Has a minimum life expectancy of 12 weeks at Screening.
* Has a left ventricular ejection fraction ≥50% within 28 days before enrollment.
* Has adequate organ and bone marrow function within 28 days before enrollment.
* Has adequate treatment washout period before enrollment.
* Male and female subjects of reproductive/childbearing potential must agree to use a highly effective form of contraception.

Exclusion Criteria:

* Prior treatment with an antibody drug conjugate (ADC).
* Uncontrolled or significant cardiovascular disease.
* Has a corrected QT interval prolongation.
* Has a history of (non-infectious) interstitial lung disease (ILD)/pneumonitis that required steroids, has current ILD/pneumonitis, or where suspected ILD/pneumonitis cannot be ruled out by imaging at Screening.
* Has spinal cord compression or clinically active central nervous system metastases.
* Has multiple primary malignancies within 3 years, except adequately resected non-melanoma skin cancer, curatively treated in situ disease, other solid tumors curatively treated, or contralateral BC.
* Has a history of severe hypersensitivity reactions to either the drug substances or inactive ingredients in the drug product.
* Has a history of severe hypersensitivity reactions to other monoclonal antibodies.
* Has an uncontrolled infection requiring intravenous (IV) antibiotics, antivirals, or antifungals.
* Active primary immunodeficiency, known uncontrolled active human immunodeficiency virus (HIV) infection, or active hepatitis B or C infection.
* Has history of receiving a live, attenuated vaccine (messenger RNA and replication-deficient adenoviral vaccines are not considered attenuated live vaccines) within 30 days prior to the first exposure to study drug.
* Has unresolved toxicities from previous anticancer therapy, defined as toxicities (other than alopecia) not yet resolved to Grade ≤1 or baseline.
* Is pregnant or breastfeeding or planning to become pregnant.
* Lung-specific intercurrent clinically significant illnesses.
* Any autoimmune, connective tissue, or inflammatory disorders.
* Prior complete pneumonectomy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2023-12-30 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Time From the Start of T-DXd to Initiation of Subsequent Anticancer Treatment (TTNT) | Until subsequent therapy or death, assessed up to 24 months
  TTNT is defined as the time interval from the date of first dose of T-DXd to the initiation of the next anticancer treatment or death due to any cause.

SECONDARY OUTCOMES:
Real-World Progression Free Survival (PFS) | Until progression or death, assessed up to 24 months
  Real-world PFS is defined as time from date of first dose of T-DXd to time of disease progression per investigator assessment based on Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 or death due to any cause.
Time From Start of T-DXd to Discontinuation of T-DXd or Death (TTD) | Until treatment discontinuation or death, up to 24 months
  TTD is defined as the time interval from the date of first dose of T-DXd to the date of discontinuation of T-DXd or death due to any cause.
Objective Response Rate (ORR) | Until progression, assessed up to 24 months
  ORR is defined as the proportion of participants with a best overall response (BOR) of confirmed complete response (CR) or confirmed partial response (PR) according to the investigator and per RECIST version 1.1 criteria.
Number of Participants With Treatment-emergent Adverse Events (TEAEs) | Up to follow up period, up to 24 months
  TEAEs are graded according to National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) v5.0. A TEAE is defined as an adverse event (AE) that occurs, having been absent before the first dose of study drug, or has worsened in severity or seriousness after initiating the study drug until 47 days after the last dose of the study drug.
Mean Change from Baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaires (EORTC-QLQ)-C30 Score | Assessed up to 24 months
  Change from baseline in the EORTC-QLQ-C30 scale scores range from 0-100. For functioning and global health status/ QoL scales, higher scores indicate better functioning or global health status/QoL. For symptom scales, higher scores indicate greater symptom burden.
Mean Change from Baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaires (EORTC-QLQ)-BR45 Score | Assessed up to 24 months
  Change from baseline in the EORTC QLQ-BR45 scale scores range from 0-100. For functioning and global health status/ QoL scales, higher scores indicate better functioning or global health status/QoL. For symptom scales, higher scores indicate greater symptom burden.
Time to First and Definitive Deterioration in European Organization for Research and Treatment of Cancer Quality of Life Questionnaires (EORTC-QLQ) Scales | Assessed up to 24 months
  Time to first and definitive deterioration in EORTC-QLQ scales. Scale scores range from 0-100. For functioning and global health status/ QoL scales, higher scores indicate better functioning or global health status/QoL. For symptom scales, higher scores indicate greater symptom burden.
Mean Change from Baseline in EuroQol Questionnaire-5 Dimensions-5 Levels (EQ-5D-5L) | Assessed up to 24 months
  Change from baseline in EQ-5D-5L. The EQ-5D-5L is a health-related QoL questionnaire based on five dimensions of health: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension contains five levels: no problems, slight, moderate, severe, and extreme problems. The EQ-5D-5L results can be converted into a single utility value. Utility values range from 0 to 1, with 1 corresponding to perfect health and 0 corresponding to a health status equivalent to death. In addition, participants can provide an overall rating of their current health status using a visual analog scale ranging from 0 (worse) to 100 (better).
Mean Change From Baseline in EuroQol Questionnaire-5 Dimensions-5 Levels (EQ-5D-5L) Index Score | Assessed up to 24 months
  Change from baseline in EQ-5D-5L index score. The EQ-5D-5L index score ranges from less than 0 (worse) to 1 (better), with higher scores representing a better health status.
Mean Change From Baseline in EuroQol Questionnaire-5 Dimensions-5 Levels (EQ-5D-5L) Visual Analog Scale (VAS) | Assessed up to 24 months
  Change from baseline in EQ-5D-5L VAS. The EQ-5D-5L VAS ranging from 0 (worse) to 100 (better) is used to assess an overall rating of participant's current health status. Higher scores indicate better clinical outcomes.
Time to First and Definitive Deterioration in EuroQol Questionnaire-5 Dimensions-5 Levels (EQ-5D-5L) Visual Analog Scale (VAS) | Assessed up to 24 months
  Time to first and definitive deterioration in EQ-5D-5L VAS. The EQ-5D-5L VAS ranging from 0 (worse) to 100 (better) is used to assess an overall rating of participant's current health status. Higher scores indicate better clinical outcomes.
Patient's Global Impression of Change (PGI-C) Response | Assessed up to 24 months
  The PGI-C is a single-item questionnaire asking for the participant's overall impression of changes in clinical condition from baseline (prior to study drug initiation), where 1 is "Normal" and 7 is "Severely ill". Lower scores indicate better clinical outcome.
Patient's Global Impression of Severity (PGI-S) Response | Assessed up to 24 months
  The PGI-S is a single-item questionnaire asking for the subject's overall impression of symptoms assessed over the past week, where 1 is "Normal" and 4 is "Severe". Lower scores indicate better clinical outcome.
Patient's Global Impression of Treatment Tolerability (PGI-TT) Response | Assessed up to 24 months
  The PGI-TT is a single-item questionnaire asking for the subject's overall impression of treatment tolerability over the past week, where 1 is "Not at all" and 5 is "Very much". Higher scores indicate a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (86):
- United States (5):
  - Mount Sinai Medical Center, Miami Beach, Florida
  - USF College of Medicine, Tampa, Florida
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Lahey Health, Burlington, Massachusetts
  - Overlook Medical Center, Summit, New Jersey
- Australia (4):
  - Mater Hospital Sydney, North Sydney, New South Wales
  - Monash Medical Centre Moorabbin, East Bentleigh, Victoria
  - GenesisCare St Andrews Hospital, Adelaide
  - Fiona Stanley Hospital, Murdoch
- Belgium (7):
  - Institut Jules Bordet, Anderlecht
  - GZA Ziekenhuizen, Antwerp
  - Universitair Ziekenhuis Brussel, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
  - UZ Leuven, Leuven
  - Centre Hospitalier Universitaire de Liege Sart-Tilman, Liège
  - GZA Ziekenhuizen, Wilrijk
- Brazil (15):
  - Centro de Oncologia - Unidade Brasília - Hospital Sírio Libanês, Brasília
  - CIONC-Centro Integrado de Oncologia de Curitiba, Curitiba
  - Hospital Erasto Gaertner - Liga Paranaense de Combate ao Câncer, Curitiba
  - CEPON - Centro de Pesquisas Oncológicas de Santa Catarina, Florianópolis
  - Oncosite - Centro de Pesquisa Clinica e Oncologia, Ijuí
  - Fundação Doutor Amaral Carvalho, Jaú
  - Instituto de Cancer de Londrina, Londrina
  - Hospital das Clínicas FMRP-USP, Riberão Preto
  - Hospital Nossa Senhora da Conceicao, Rio Grande
  - Ensino e Terapia de Inovação Clínica AMO-ETICA, Salvador
  - Catarina Pesquisa Clinica, Santa Catarina
  - CEPHO - Centro de Estudos e Pesquisas de Hematologia e Oncologia, Santo André
  - Fundacao Faculdade Regional de Medicina de Sao Jose do Rio Preto, São José do Rio Preto
  - ICESP - Instituto do Câncer do Estado de São Paulo Octavio Frias de Oliveira, São Paulo
  - Clínica de Pesquisas e Centro de Estudos em Oncologia Ginecológica e Mamária Ltda, São Paulo
- China (13):
  - Beijing Hospital, Beijing
  - 307 Hospital of PLA, Beijing
  - Fujian Cancer Hospital, Fujian
  - Sun Yat sen University Cancer Center, Guangzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - Anhui Provincial Cancer Hospital, Hefei
  - Shandong Cancer Hospital, Jinan
  - Yunnan Cancer Hospital, Kunming
  - Nanchang People's Hospital, Nanchang
  - Jiangxi Cancer Hospital, Nanchang
  - The Affiliated Hospital of Qingdao University, Qingdao
  - Fudan University Shanghai Cancer Center, Shanghai
  - Henan Cancer Hospital, Zhengzhou
- Ireland (5):
  - Cork University Hospital, Cork
  - St Vincent's University Hospital, Dublin
  - St James Hospital, Dublin
  - Beaumont Hospital, Dublin
  - Galway University Hospital, Galway
- Italy (11):
  - Istituto Tumori Giovanni Paolo II IRCCS Ospedale Oncologico Bari, Bari
  - Azienda Ospedaliera Universitaria Policlinico Sant Orsola Malpighi IRCCS, Bologna
  - Istituto Nazionale per la Ricerca sul Cancro di Genova, Genova
  - Ospedale San Raffaele, Milan
  - Humanitas Istituto Clinico Catanese, Misterbianco
  - Istituto Nazionale Tumori Fondazione G Pascale, Naples
  - IOV - Istituto Oncologico Veneto IRCCS, Padua
  - Nuovo Ospedale di Prato, Prato
  - Azienda Ospedaliera Universitaria Policlinico Umberto I - Università di Roma La Sapienza, Rome
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome
  - Ospedale Santa Chiara, Trento
- Netherlands (8):
  - Amsterdam UMC, Locatie VUMC, Amsterdam
  - Amphia Ziekenhuis Molengracht, Breda
  - Medisch Centrum Leeuwarden, Leeuwarden
  - Alrijne Ziekenhuis Leiden, Leiden
  - Maastricht University Medical Center, Maastricht
  - Haga Ziekenhuis, The Hague
  - Elisabeth TweeSteden Ziekenhuis, Tilburg
  - Bernhoven Uden, Uden
- Portugal (4):
  - Hospital de Braga, Braga
  - Instituto Português de Oncologia de Lisboa Francisco Gentil, EPE, Lisbon
  - Fundação Champalimaud, Lisbon
  - Centro Hospitalar de Lisboa Norte E P E Hospital de Santa Maria, Lisbon
- Spain (14):
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - ICO l'Hospitalet - Hospital Duran i Reynals, Barcelona
  - Hospital Universitario Donostia, Donostia / San Sebastian
  - Hospital Universitario Virgen de las Nieves, Granada
  - Complejo Hospitalario Universitario Insular Materno-Infantil, Las Palmas de Gran Canaria
  - Hospital Beata Maria Ana, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda
  - Hospital General Universitario Morales Meseguer, Murcia
  - Clinica Universidad de Navarra, Pamplona
  - Complejo Hospitalario Universitario de Santiago, Santiago de Compostela
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Clinico Universitario de Valencia, Valencia
  - Hospital Arnau de Vilanova de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) on completed studies and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Completed studies that has reached a global end or completion with all data set collected and analyzed, and for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents on completed clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- [Derived] Yaziji H, Hornick JL, Troxell ML. The Suitability of Repurposed, Legacy HER2 Immunohistochemistry Assays for the Detection of HER2 Low and Ultralow Expression: Current Limitations and Potential Considerations. Appl Immunohistochem Mol Morphol. 2026 Jan 1;34(1):1-4. doi: 10.1097/PAI.0000000000001296. Epub 2025 Dec 4. No abstract available. PMID 41342740